CLINICAL TRIAL: NCT06448130
Title: Effect of Henagliflozin on the Remission of Prediabetes Population: A National Multicenter, Randomized Controlled Study
Brief Title: Henagliflozin's Impact on Prediabetes Remission
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Jia-jun Zhao, Principal Investigator, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MA-DM-IV-004
Record Dates: First submitted 2024-05-15; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: PreDiabetes; Prediabetic State; Type 2 Diabetes; Glucose Metabolism Disorders
Keywords: Prediabetes management; Henagliflozin; SGLT2 inhibitors; Lifestyle interventions; Type 2 diabetes prevention; Glucose Metabolism Disorders; Metabolic Diseases
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases | interventions — henagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Henagliflozin5mg + lifestyle intervention (Experimental): Henagliflozin 5mg+ placebo 10mg po qd + lifestyle intervention for 6 months
  Interventions: Drug: Henagliflozin 5mg
- Henagliflozin10mg+ lifestyle intervention (Experimental): Henagliflozin 10mg+ placebo 5mg po qd + lifestyle intervention for 6 months
  Interventions: Drug: Henagliflozin 10mg
- placebo+ lifestyle intervention (Placebo Comparator): placebo 10mg + placebo 5mg po qd + lifestyle intervention for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Henagliflozin 5mg — Henagliflozin 5mg + lifestyle intervention
  Other Names: lifestyle intervention
  Arms: Henagliflozin5mg + lifestyle intervention
Drug: Henagliflozin 10mg — Henagliflozin 10mg+ lifestyle intervention
  Other Names: lifestyle intervention
  Arms: Henagliflozin10mg+ lifestyle intervention
Drug: Placebo — Placebo+ lifestyle intervention
  Other Names: lifestyle intervention
  Arms: placebo+ lifestyle intervention

SUMMARY:
This clinical trial evaluates the effectiveness of Henagliflozin combined with lifestyle interventions for managing patients with prediabetes. As global prediabetes rates rise, increasing the risk of diabetes and vascular issues, addressing treatment gaps is essential. Henagliflozin, a novel SGLT2 inhibitor developed in China, aims to improve glucose control and metabolic health when paired with lifestyle changes.

The study's primary objectives include: assessing whether Henagliflozin can achieve normoglycemia in prediabetic patients after 6 months of treatment.

The trial will compare three groups (Henagliflozin 5mg, 10mg, and a placebo), focusing on efficacy and safety. Participants, assigned randomly, will undergo a 6-month treatment phase and an 18-month follow-up. Regular health assessments will monitor glucose levels, metabolic health, and risks of major complications like cardiovascular events and microvascular diseases, with additional evaluations of C-peptide and insulin changes.

Structured as a multicenter, randomized, double-blind, placebo-controlled study, it involves 984 prediabetic adults across 50 medical institutions in China. This comprehensive approach could redefine prediabetes management by integrating drug therapy with lifestyle modifications.

DETAILED DESCRIPTION:
This research is launched in light of the global surge in prediabetes, a condition that markedly increases the risk of developing type 2 diabetes and related vascular complications. While lifestyle modifications are the frontline defense against prediabetes, the variability in individual responses often requires the integration of pharmacological treatments. Studies have shown that drugs such as metformin, acarbose, SGLT2 inhibitors, GLP-1 agonists, GIP/GLP-1 receptor agonists, thiazolidinediones, and orlistat effectively curb the progression to diabetes. Yet, there remains a gap in specific research addressing the intervention needs of the prediabetic population in China.

Currently, acarbose is the only drug approved in the Chinese market for treating patients with impaired glucose tolerance, highlighting a limited range of therapeutic options for prediabetes. SGLT2 inhibitors, as a newer class of hypoglycemic agents, have demonstrated significant promise in reducing major cardiovascular events in high-risk patients with type 2 diabetes, enhancing outcomes in heart failure, and providing renal protection. However, there is a scarcity of large-scale, prospective studies on the impact of SGLT2 inhibitors in prediabetes. Henagliflozin, the first original SGLT2 inhibitor developed in China and launched on December 31, 2021, is being studied to assess its effectiveness combined with lifestyle interventions in the prediabetic demographic, aiming to fill a crucial void in the current treatment paradigm.

This study aims to assess the combined benefits of Henagliflozin and lifestyle modifications in managing prediabetes. The investigators conducted a two-year prospective, randomized, double-blind, placebo-controlled trial across 50 medical institutions in various provinces of China. It is planned to enroll 984 adult prediabetic patients who had not previously been treated with antidiabetic medications. Participants meeting inclusion criteria were randomly assigned to one of three groups: Henagliflozin 5mg, Henagliflozin 10mg, or placebo. The intensive intervention phase, consisting of pharmacotherapy combined with lifestyle changes, lasted for 6 months, followed by an 18-month follow-up period focusing solely on lifestyle interventions.

The primary endpoint is the proportion of participants achieving normoglycemia after 6 months of intervention, with subsequent assessments at 12 months. Secondary endpoints include short-term (0-12 months) and long-term (12-24 months) changes in glucose control, metabolic indicators such as body weight, body mass index (BMI), body fat content, waist and hip circumference, lipid profiles, blood pressure, serum uric acid levels, hepatic steatosis, and carotid intima-media thickness. Exploratory outcomes encompass changes in C-peptide and insulin levels from baseline to 6 months, and the risk of major adverse cardiovascular events (MACE) from baseline to 24 months and beyond.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between the ages of 18 and 65 years;
2. Individuals without hypoglycemic therapy before, including hypoglycemic drugs or traditional Chinese medicine formulations with hypoglycemic effects;
3. Prediabetic patients as defined by Expert Consensus on Intervention for Prediabetes in Chinese Adults, 2023 Edition:1)Fasting plasma glucose (FPG) between 6.1 and 7.0 mmol/L and/or 2-hour postprandial glucose (2h-PPG) between 7.8 and 11.1 mmol/L; 2)And/or HbA1c between 5.7% and 6.5%;
4. Individuals willing to provide written informed consent and can comply with study procedures and follow-up.

Exclusion Criteria:

1. Allergic to Henagliflozin;
2. Previously diagnosed with diabetes;
3. HbA1c ≥ 6.5% or FPG ≥ 7.0 mmol/L or PPG ≥ 11.1 mmol/L;
4. Use of GLP-1 receptor agonists, orlistat, or other weight-reducing drugs in the past 3 months;
5. Fluctuation in weight by 5% or more in the past month;
6. Use of drugs affecting glucose synthesis, absorption, or metabolism, such as glucocorticoids (e.g., prednisone, dexamethasone), contraceptives, growth hormone, hormonal replacement therapy (estrogen and progesterone), immunosuppressants (e.g., cyclosporine A, tacrolimus), anti-tuberculosis drugs (e.g., isoniazid, rifampicin);
7. Untreated hyperthyroidism or hypothyroidism, excluding those with normal thyroid function after treatment;
8. Persistently uncontrolled hypertension (used antihypertensive drugs but was not effectively controlled in the 3 months prior to enrollment) or currently use 3 or more antihypertensive drugs (including diuretics);
9. Assessed by the investigator to be at high risk of genitourinary system infections, such as history of recurrent urinary tract infections or reproductive system infections, long-term placement of urinary catheters, or history of urological surgery;
10. Other obesity caused by endocrine disorders, such as Cushing's syndrome;
11. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels > 3 times of the upper limit of the normal range (UNL);
12. eGFR less than 30 mL/min/1.73 m2, severe kidney damage, end-stage renal disease or requiring dialysis;
13. Significant cardiovascular diseases including myocardial infarction, congestive heart failure (≥grade III New York Heart Association), left ventricular ejection fraction≤40%, or cerebrovascular accidents;
14. Impaired consciousness and various mental health disorders;
15. Malignant tumors and other serious illnesses;
16. Pregnant or breast-feeding or planning pregnancy within 24 months;
17. Enrolled in another clinical trial currently or within the 3 months prior to enrollment;
18. Identified by the investigator that lacks sufficient motivation to continue the long-term clinical trial (e.g., out-of-town study, work plan, need to care for family members), or considered prefer to withdraw from the trial for non-medical reasons (such as social issues).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 984 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Normoglycemia Achievement Rates Post-6-Month Intervention | From 6 months post-intervention to 12 months
  This measure assesses the proportion of participants who achieve normoglycemia from the end of a 6-month intervention until the 12-month assessment point. Normoglycemia is defined as fasting plasma glucose (FPG) less than 6.1 mmol/L and 2-hour post-prandial glucose (2h-PPG) less than 7.8 mmol/L. The measure includes rates of sustained remission (normal glycemic status lasting more than 6 months post-medication cessation), partial remission (lasting 3-6 months), and temporary remission (lasting less than 3 months).

SECONDARY OUTCOMES:
Blood Glucose Control Normalization | From 6 months post-intervention to 24 months
  Proportion and duration of normalization of blood glucose levels within 24 months in the three study groups.
Incidence of New-Onset Type 2 Diabetes | From 0 to 24 months
  Incidence of new-onset type 2 diabetes within 24 months in the three study groups.
Changes in HbA1c Levels | From 0 to 24 months
  Changes in HbA1c levels over the 24-month period in the three study groups.
Impact of Glycemic Status at 12 Months | From 12 months to 24 months
  Impact of glycemic status at 12 months on subsequent reversal to normoglycemia and risk of new-onset type 2 diabetes during the 12-24 month follow-up period in the three study groups.
Changes in blood pressure over 24 Months | From 0 to 24 months
  Changes in systolic and diastolic blood pressure in the three study groups over 24 Months.
Changes in serum uric acid levels over 24 Months | From 0 to 24 months
  Changes in serum uric acid levels in the three study groups over 24 Months.
Changes in hepatic steatosis over 24 Months | From 0 to 24 months
  Changes in hepatic steatosis assessed by abdominal ultrasound in the three study groups over 24 Months.
Changes in carotid intima-media thickness over 24 Months | From 0 to 24 months
  Changes in carotid intima-media thickness measured by carotid ultrasound in the three study groups over 24 Months.
Changes in Total Cholesterol (TC) over 24 Months | From 0 to 24 months
  Measurement of Total Cholesterol (TC) levels in millimoles per liter (mmol/L) using standardized laboratory procedures. Fasting blood samples will be collected at multiple time points within the 24-month period to assess changes over time.
Changes in Triglycerides (TG) over 24 Months | From 0 to 24 months
  Measurement of Triglycerides (TG) levels in millimoles per liter (mmol/L) using standardized laboratory procedures. Fasting blood samples will be collected at multiple time points within the 24-month period to assess changes over time.
Changes in Low-Density Lipoprotein Cholesterol (LDL-c) over 24 Month | From 0 to 24 months
  Measurement of Low-Density Lipoprotein Cholesterol (LDL-c) levels in millimoles per liter (mmol/L) using standardized laboratory procedures. Fasting blood samples will be collected at multiple time points within the 24-month period to assess changes over time.
Changes in High-Density Lipoprotein Cholesterol (HDL-c) over 24 Months | From 0 to 24 months
  Measurement of High-Density Lipoprotein Cholesterol (HDL-c) levels in millimoles per liter (mmol/L) using standardized laboratory procedures. Fasting blood samples will be collected at multiple time points within the 24-month period to assess changes over time.
Changes in Body Weight over 24 Months | From 0 to 24 months
  Measurement of body weight in kilograms (kg) at multiple time points within the 24-month period.
Changes in Body Mass Index (BMI) over 24 Months | From 0 to 24 months
  Calculation of BMI in kg/m² using the formula: weight (kg) / (height (m)²), measured at multiple time points within the 24-month period.
Changes in Body Fat Content over 24 Months | From 0 to 24 months
  Measurement of body fat content as a percentage (%) of total body weight at multiple time points within the 24-month period.
Changes in Waist Circumference over 24 Months | From 0 to 24 months
  Measurement of waist circumference in centimeters (cm) at multiple time points within the 24-month period.
Changes in Hip Circumference over 24 Months | From 0 to 24 months
  Measurement of hip circumference in centimeters (cm) at multiple time points within the 24-month period.
Changes in C-peptide Levels over the First 6 Months | From 0 to 6 months
  Measurement of C-peptide levels in nanomoles per liter (nmol/L) at multiple time points within the 6-month period.
Changes in Insulin Levels over the First 6 Months | From 0 to 6 months
  Measurement of insulin levels in milliunits per liter (mU/L) at multiple time points within the 6-month period.
Major Adverse Cardiovascular Events | From 0 to 24 months
  Major Adverse Cardiovascular Events (MACE) in the three study groups over 0-24 months.
Risk of Retinal Diseases | From 0 to 24 months
  Risk of retinal diseases (e.g., diabetic retinopathy) in the three study groups over 0-24 months.
Risk of Renal diseases | From 0 to 24 months
  Risk of renal diseases (e.g., diabetic nephropathy/chronic kidney disease) in the three study groups over 0-24 months.

CONTACTS AND LOCATIONS:
Locations (50):
- China (50):
  - Chuzhou First People's Hospital, Chuzhou, Anhui
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - LanZhou University, Lanzhou, Gansu
  - Shunde Hospital of Southern Medical University, Foshan, Guangdong
  - Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guanzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - North China University of Technology Affiliated Hospital, Tangshan, Hebei
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Xinyang Central Hospital, Xinyang, Henan
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Second Affiliated Hospital of Nanchang University, Nanchang, Jiangsu
  - The First Affiliated Hospital with Nanjing Medical University,, Nanjing, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - People's Hospital of Liaoning Province, Shenyang, Liaoning
  - Ningxia Medical University, Yinchuan, Ningxia
  - Binzhou City Central Hospital, Binzhou, Shandong
  - Dongying People's Hospital, Dongying, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - The Second Affiliated Hospital of Shandong First Medical University, Tai’an, Shandong
  - The Affiliated Hospital of Weifang Medical University, Weifang, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Yantai Affiliated Hospital of Binzhou Medical University, Yantai, Shandong
  - Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Central Hospital of Lishui City, Lishui, Zhejiang
  - First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Wenzhou Central Hospital, Wenzhou, Zhejiang
  - Beijing Hospital, Beijing
  - Beijing Luhe Hospital, Beijing
  - Beijing Chao Yang Hospital, Beijing
  - First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Baoshan Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai
  - Shanghai 10th People's Hospital, Shanghai
  - Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University, Shanghai
  - Peking University Binhai Hospital, Tianjin
  - Tianjin First Central Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Undecided
We have opted for 'Undecided' regarding the sharing of individual participant data (IPD) at this stage. Our decision is pending as we are currently engaged in ongoing discussions and evaluations regarding the most appropriate approach to IPD sharing for our research. Factors such as ethical considerations, data sensitivity, and regulatory requirements are being carefully assessed. We aim to reach a well-informed decision in due course and will update our IPD sharing plan accordingly. Thank you for your understanding as we navigate through this process.